CLINICAL TRIAL: NCT05075096
Title: Long Term Outcome in ICU Treated COVID-19: New Chronic Diseases
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Dalarna County Council, Sweden (Other)
Responsible Party: Sponsor
Other Study IDs: U1111-1269-6916
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Covid19
Keywords: Long term outcome; Mortality; COVID-19; Morbidity
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COVID-19 ICU cohort: All patients admitted to a Swedish ICU with COVID-19 with at least one year of follow up. COVID-19 defined by the ICD-10 diagnosis U07.1 in the nationwide Swedish intensive care registry.
  Interventions: Other: No intervention.
- COVID-19 hospital admission control cohort: Four random control patients per ICU patient matched on age legal gender and region. Controls selected from all patients admitted to a Swedish hospital with COVID-19 with at least one year of follow up. Not including patients in the COVID-19 ICU cohort. COVID-19 defined by the ICD-10 diagnosis U07.1 in the nationwide Swedish national patient registry.
  Interventions: Other: No intervention.
- General population control cohort: Four general population controls per ICU patient, matched on age, legal gender and region drawn from the total population register of Sweden. Not including ICU and hospital admitted COVID-19 patients.
  Interventions: Other: No intervention.

INTERVENTIONS:
Other: No intervention. — No intervention observational study.

SUMMARY:
Additional chronic diseases one year after intensive care unit (ICU) admission with Coronavirus disease 2019 (COVID-19) will be assessed in comparison to two control cohorts.

The ICU population comprises all Swedish ICU patients with COVID-19 with at least one year of follow up. The hospital admitted cohort comprises four hospital admitted patients with COVID-19 per ICU patient, matched on age, legal gender and region. The general population controls are matched to the ICU patients in a one to four fashion on age, legal gender and region.

ICU patients are identified in the Swedish intensive care registry. The hospital admitted patients are identified in the national patient registry and the population controls are identified in the population registry. Data on comorbidity, medications and death are provided from the National board of health and welfare.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to a Swedish ICU and registered in the Swedish intensive care registry with the ICD 10 diagnosis U07.1 before 1 July 2020. ICU-cohort.

or randomly selected from all patients admitted to hospital but not ICU with the ICD 10 diagnosis U07.1 in the national patient registry, matched on age, legal gender and region (four per ICU patient) before 1 July 2020. Hospital cohort.

or randomly selected from the general population (and not included in the ICU or hospital admitted cohorts), matched on age, legal gender and region (four per ICU patient)

Exclusion Criteria:

* Missing a Swedish personal identification number

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of all patients a fulfilling the eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 60000 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Is the illness severity in COVID-19 (according to level of care cohort) an independent risk factor for incident chronic renal failure within one year after inclusion? | One year
  Variables in binary logistic model with the outcome incident chronic renal failure: On sick leave one year before ICU admission, age, legal gender, highest education, immigrant background, income the year before inclusion, marital status co-morbid diabetes mellitus. Interaction with a variable denoting cohort (ICU, Hospital or General population) is added to all variables. A significant interaction indicates a differential effect between cohorts.
Is the illness severity in COVID-19 (according to level of care cohort) an independent risk factor for incident pulmonary disease within one year after inclusion? | One year
  Variables in binary logistic model with the outcome incident pulmonary disease: On sick leave one year before ICU admission, age, legal gender, highest education, immigrant background, income the year before inclusion, marital status. Interaction with a variable denoting cohort (ICU, Hospital or General population) is added to all variables. A significant interaction indicates a differential effect between cohorts.
Is the illness severity in COVID-19 (according to level of care cohort) an independent risk factor for incident cardiac failure within one year after inclusion? | One year
  Variables in binary logistic model with the outcome incident cardiac failure: On sick leave one year before ICU admission, age, legal gender, highest education, immigrant background, income the year before inclusion, marital status co-morbid ischemic heart disease. Interaction with a variable denoting cohort (ICU, Hospital or General population) is added to all variables. A significant interaction indicates a differential effect between cohorts.
Is the illness severity in COVID-19 (according to level of care cohort) an independent risk factor for incident pulmonary hypertension within one year after inclusion? | One year
  Variables in binary logistic model with the outcome incident pulmonary hypertension: On sick leave one year before ICU admission, age, legal gender, highest education, immigrant background, income the year before inclusion, marital status co-morbid chronic obstructive pulmonary disease. Interaction with a variable denoting cohort (ICU, Hospital or General population) is added to all variables. A significant interaction indicates a differential effect between cohorts.
Is the illness severity in COVID-19 (according to level of care cohort) an independent risk factor for being diagnosed with Post COVID (ICD-10, U09.9) within one year after inclusion? | One year
  Variables in binary logistic model with the outcome Post COVID: On sick leave one year before ICU admission, age, legal gender, highest education, immigrant background, income the year before inclusion, marital status. Interaction with a variable denoting cohort (ICU, Hospital or General population) is added to all variables. A significant interaction indicates a differential effect between cohorts.
Is the illness severity in COVID-19 (according to level of care cohort) an independent risk factor for incident psychiatric disease within one year after inclusion? | One year
  Variables in binary logistic model with the outcome incident psychiatric disease: On sick leave one year before ICU admission, age, legal gender, highest education, immigrant background, income the year before inclusion, marital status. Interaction with a variable denoting cohort (ICU, Hospital or General population) is added to all variables. A significant interaction indicates a differential effect between cohorts.

SECONDARY OUTCOMES:
Is the prevalence of pulmonary disease, chronic renal failure, pulmonary hypertension, cardiac failure or psychiatric diseases more common one year after than before ICU admission with COVID-19? | One year
  Analyzed in the ICU admitted cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Miklos Lipcsey, Professor, Principal Investigator — 202100-2932
Locations (1):
- Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No
IPD sharing is not allowed under the ethical review approval.